CLINICAL TRIAL: NCT07190404
Title: Efficacy and Mechanisms of a Metacognitive Strategy Intervention for Parkinson Disease-Related Cognitive Decline.
Brief Title: Multicontext Approach for Cognitive Function in Parkinson Disease
Acronym: MC4PD R01
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Erin Foster, Associate Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202508056
Record Dates: First submitted 2025-09-09; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: Parkinson Disease; occupational therapy
MeSH Terms: conditions — Parkinson Disease | interventions — Microscopy, Electron, Scanning Transmission

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MC Approach (Experimental): The experimental Multicontext Approach Intervention
  Interventions: Behavioral: A metacognitive strategy for cognitive rehabilitation called the Multicontext Approach.
- Process Training (Active Comparator): The Control Group cognitive process training
  Interventions: Behavioral: Cognitive (Process) Training
- MC + Booster (Experimental): From the MC Approach group only, MC+Boster participants will receive 2 additional treatment sessions with their original OT within the month following their 6mo FU assessment.
  Interventions: Behavioral: MC Approach Booster Session

INTERVENTIONS:
Behavioral: A metacognitive strategy for cognitive rehabilitation called the Multicontext Approach. — The Multicontext Approach is a strategy training approach to cognitive intervention provides ways to maintain daily function despite the presence of cognitive deficits. It involves teaching people to use metacognitive, compensatory, or adaptive techniques to optimize information processing or bypass cognitive limitations and achieve task-related goals. Strategy training is recommended for those with mild (vs. more severe) cognitive deficits because it requires learning, capitalizes on existing cognitive resources, and aims to prevent or delay functional decline.
  Arms: MC Approach
Behavioral: Cognitive (Process) Training — This treatment is functional task training, a widely-used approach in neurorehabilitation153,154 that parallels the cognitive training used in PD to-date but with functional cognitive tasks (vs. computer or paper & pencil tasks) to improve ecological validity. It has the same structure within and across treatment sessions and uses the same treatment activities as the MC intervention. However, the OT does not use mediated learning techniques or explicitly address strategies, metacognition, or transfer/generalization. Rather, participants practice functional cognitive tasks with knowledge of results feedback and cueing by the OT to improve task performance.
  Arms: Process Training
Behavioral: MC Approach Booster Session — MC+B participants will come from the MC Approach group only. They will receive 2 additional treatment sessions with their original OT within the month following their 6mo FU assessment. The OT will review the participant's relevant Post and FU data beforehand for treatment planning purposes. The first session will involve a review of goals, prior learning, and strategies and discussion of successes/challenges related to functional cognitive performance and strategy application since initial treatment. Then the same protocol (treatment activities with metacognitive framework and mediation, strategy bridging discussions, homework action planning and review) will be followed for the rest of the booster treatment to reinforce or re-activate prior learning, address new concerns, and develop supports for maintenance.
  Arms: MC + Booster

SUMMARY:
Mild cognitive decline is common in early Parkinson disease (PD) and is associated with disability, reduced quality of life (QOL), and increased risk for dementia. Medical treatments for PD do not prevent or treat cognitive decline and may even exacerbate the problem.

Unfortunately, existing cognitive interventions for PD, which focus on restoring deficient cognitive skills through cognitive training (repetitive practice of tasks that challenge specific cognitive skills), provide limited benefit for daily function and QOL. To overcome this limitation, the investigators use strategy training. the investigators help people develop targeted strategies to use in everyday life to circumvent cognitive deficits and accomplish daily activities. Contemporary cognitive rehabilitation evidence supports strategy training for other neurological conditions and mild cognitive impairment (MCI), but it has not been well-studied in PD. By teaching strategies for everyday cognition, the investigators hypothesize that our interventions will improve functional outcomes for people with PD.

Study participants will complete a baseline cognitive testing session, 10 cognitive treatment sessions with a trained occupational therapist, then have follow-up visits with the study team at 1-week, 3-months, 6-months, and 12-months after completing the study intervention.

DETAILED DESCRIPTION:
Mild cognitive decline is common in early Parkinson disease (PD) and is associated with disability, reduced quality of life (QOL), and increased risk for dementia. Medical treatments for PD do not prevent or treat cognitive decline and may even exacerbate the problem. Therefore, behavioral interventions that attenuate its negative functional consequences and thus potentially delay dementia onset are a top research priority. Unfortunately, existing cognitive interventions for PD, which focus on restoring deficient cognitive skills through cognitive training (repetitive practice of tasks that challenge specific cognitive skills), provide limited benefit for daily function and QOL. To overcome this limitation, the investigators use strategy training. the investigators help people develop targeted strategies to use in everyday life to circumvent cognitive deficits and accomplish daily activities. Contemporary cognitive rehabilitation evidence supports strategy training for other neurological conditions and mild cognitive impairment (MCI), but it has not been well-studied in PD. By teaching strategies for everyday cognition, the investigators hypothesize that our interventions will improve functional outcomes for people with PD.

Specifically, the investigators use the Multicontext (MC) Approach to support daily cognitive function in people with PD with mild cognitive decline. The MC Approach is a metacognitive strategy intervention that targets awareness, strategy use, and self-efficacy to improve functional cognitive performance in daily life. Through therapist- mediated experiences with cognitively challenging functional activities, participants develop personalized strategies (e.g., self-talk, planning, checklists) to prevent or correct cognitive performance errors. The goal is to enable people to manage everyday cognitive challenges so they can perform and participate in meaningful activities and roles. In a development and proof-of-concept study, the investigators adapted and refined the treatment protocol and training materials, established good participant acceptance, and provided preliminary data on its benefits for daily cognitive function. In a subsequent pilot quasi-randomized controlled trial (R21AG063974), the investigators established trial feasibility and treatment fidelity and generated promising treatment effect data. Notably, the MC Approach produced clinically meaningful improvements in daily cognitive function that were larger than that of the cognitive task training control and that were maintained 3 and possibly 12 months post treatment. the investigators now have the experience, methods, and data to justify and prepare us for a full-scale efficacy trial.

The investigators will conduct a randomized controlled trial (RCT) to determine the short- and long-term efficacy of the MC Approach for improving daily cognitive function in people with PD with mild cognitive decline. Secondarily, the investigators will examine whether booster treatment enhances treatment effects and explore the cognitive-behavioral mechanisms of the MC Approach. PD participants (N=114) will complete baseline assessment, randomization to treatment group (MC n=76, Control n=38), 10 treatment sessions (1x/week), and 1 week, 3 months, and 6 months post treatment assessment. MC participants will then be randomized to a booster (MC+B n=38) or no-booster (MC n=38) condition, and the MC+B group will receive booster treatment within the following month. Then all three groups (Control, MC, MC+B) will complete 12-month assessment. Mixed model repeated measures analysis of variance will be used to compare change across treatment groups and over time.

Our primary study aims and hypotheses are:

Aim 1: Determine the effect of the MC Approach on daily cognitive function. H1: The MC group will report greater improvements in daily cognitive function than the Control group 1 week (H1a; short-term) and 12 months (H1b; long-term) post treatment. Participants will rate their performance on personalized functional cognitive goals using a standardized cognitive rehabilitation tool (primary outcome: Bangor Goal Setting Interview, (BGSI) at each testing timepoint. Primary analyses will include the 1-week and 12-month data for Control and MC participants; additional analyses can look at trajectories across all timepoints.

Aim 2: Examine the effect of booster MC Approach treatment on daily cognitive function.

H2: The MC+B group will report better daily cognitive function 12 months post initial treatment than the MC group. At 6 months post, MC+B participants will receive two booster treatment sessions to review and reinforce their learning and strategy use. Primary analyses will include the 6- and 12-month BGSI data, controlling for baseline.

Aim 3: Explore the effect of the MC Approach on the theorized intermediate treatment targets.

H3: The MC group will have greater improvements in awareness, strategy use, and self-efficacy than the Control group after treatment. Participants will complete measures of awareness, strategy use, and self-efficacy at each testing timepoint. Primary analyses will include all available timepoints. To further explore mechanisms of action, correlational analyses will examine if change in the targets relates to change in functional outcomes.

ELIGIBILITY:
Inclusion criteria:

1. Males and females over age 50 who meet criteria for typical idiopathic PD.
2. Hoehn & Yahr stage I-III.
3. Have subjective cognitive decline (SCD) as defined by a positive answer to either question:

   * Do you feel like your thinking skills or memory are becoming worse or are worse than others your age?
   * Do you have problems or concerns with your thinking skills or memory?, and can list ≥1 daily cognitive challenge they want to address.
4. Medications should be stable for 4 weeks prior with no changes planned during the treatment portion of the study (Pre to Post); unplanned changes and changes over the follow-up period will be tracked and accounted for as appropriate.

Exclusion criteria:

1. Dementia according to MDS criteria or MoCA score <21.
2. Other neurological disorders (e.g., stroke, seizures).
3. Current or history of major psychiatric disorder or psychotic symptoms (e.g., schizophrenia, bipolar disorder, delusions, hallucinations), drug abuse. Psychiatric conditions/symptoms that are common in PD (e.g., anxiety, depression) are permitted if deemed insufficient to interfere with participation.
4. Other circumstance that would interfere with participation (e.g., non-English speaking, blindness, lives >50mi away).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Bangor Goal Setting Interview | Goals will be assessed during the intervention at 2- and 4-weeks after Baseline testing; at POST intervention 11-weeks after Baseline; then one year from the final intervention session (63-weeks after Baseline).
  A standardized cognitive rehabilitation tool to identify functional cognitive problems and develop treatment goals. Participants rate their goal attainment on a scale from 0 (not successful) to 10 (very successful); readiness to work on the specific goal on a scale of 0 (not ready to change) to 10 (Extremely ready to change); and the importance of the goal to them on a scale from 0 (not important) to 10 (extremely important).

SECONDARY OUTCOMES:
The Cognitive Self-Efficacy Questionnaire | Participants will complete this questionnaire at the Baseline session, then after the participant finishes the intervention sessions at 11-, 23-, 35- and 63-weeks after Baseline.
  A self-reported questionnaire of a person's confidence in their ability to handle cognitively or mentally challenging situations. Participants rate their self-recognition of cognitive lapses (higher score indicates better recognition of cognitive lapses); their confidence to complete cognitively challenging situations (higher score indicates higher confidence); and their self-efficacy for everyday cognitive tasks (higher scores indicate higher self-efficacy).
The Weekly Calendar Planning Activity | The weekly calendar planning activity is administered at treatment session 1 of the intervention (1 week after Baseline), then after the participant completes the intervention at 11- and 63-weeks after Baseline.
  A performance-based assessment of executive function. The activity involves following and organizing a list of appointments or errands into a weekly schedule while keeping track of rules, and avoiding scheduling conflicts. Participants are scored on how many appointments are entered accurately, how many are missing or have errors (total of 17 possible). The total time it takes to complete the task is also measured. Observations are also made about any cognitive strategies used during the task.
The Self-Regulation Skills Interview | Participants are interviewed with the SRSI at treatment session 1 of the intervention (1 week after Baseline) then 1-week post intervention (11 weeks after Baseline).
  A clinical tool designed to measure a range of metacognitive skills essential for rehabilitation planning. Participants are asked in an interview what their main area of cognitive difficulty is, their awareness of this difficulty and in what situations they experience it, and if they know of any strategies or are using any strategies that they could use to cope with their main cognitive difficulty. They are also rated on their motivation to learn new strategies on a scale of 0 (Not at all) to 10 (Very motivated).

CONTACTS AND LOCATIONS:
Overall Officials: Erin R Foster, PhD, OTDR/L, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
This project will generate data obtained from participant surveys, interviews and cognitive testing, and care partner surveys. Data will be collected from 114 adults with Parkinson disease (PD) and their care partners at baseline and then 1 week, 3 months, 6 months and 12 months after treatment, generating 1 longitudinal quantitative dataset. Individual data (with identifiers removed and not linkable) will be made available for sharing. All data produced from this project will be preserved and shared to maximize the potential of knowledge gained from this dataset and the time/effort contributed by the participants. Data will be stored in common and open formats, (e.g., csv, txt, pdf, html) and deposited into Digital Commons Data@Becker, which is maintained at Bernard Becker Medical Library at WUSM.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Shared data generated from this project will be made available as soon as possible, and no later than the time of publication or within 9 months of database lock, whichever comes first. The duration of preservation and sharing of the data will be a minimum of 5 years after the end of the funding period.
Access Criteria: Human subjects' data will be shared within IRB bounds. WashU HRPO (Human Research Protection Office) typically recommends sharing de-identified data in a controlled manner. We will share de-identified data in Digital Commons@Becker, requiring requestors to sign a Data Use Agreement (DUA) unless directed otherwise by WashU HRPO/IRB.
URL: https://digitalcommons.wustl.edu/